CLINICAL TRIAL: NCT06349031
Title: Comparison of Efficacy & Tolerability Of Polyethylene Glycol 4000 Versus Polyethylene Glycol 3350+ Electrolytes For Fecal Disimpaction in Pediatric Functional Constipation: A Double-Blind Randomized Controlled Trial
Brief Title: Comparison of Efficacy & Tolerability Of PEG 4000 Versus PEG 3350+ Electrolytes for Pediatric Fecal Disimpaction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Sciences and SUM Hospital (Other)
Responsible Party: Principal Investigator, Kalpana Panda, Associate Professor, Institute of Medical Sciences and SUM Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC/IMS.SH/SOA/2024/683
Record Dates: First submitted 2024-03-30; First posted 2024-04-05 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Functional Constipation; Fecal Impaction; Constipation - Functional; Constipation Chronic Idiopathic; Pediatric Functional Constipation
Keywords: Functional constipation; Fecal disimpaction; pediatric; Polyethelene glycol 3350; Polyethylene glycol 4000
MeSH Terms: conditions — Fecal Impaction | interventions — Electrolytes

STUDY DESIGN:
Intervention Model Description: DOUBLE BLIND RANDOMIZED CONTROLLED TRIAL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One member of the research group will do the treatment allocation and will not be involved in clinical evaluation and collection of outcome data. Both study medications will be provided by him/her in opaque bottles with identical packaging and labeling. Neither the participants nor the rest of the study personnel will be aware of the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyethylene glycol (PEG) 3350 +Electrolytes ARM (Active Comparator): [PEG 33500+Electrolyte] will be administered at a dose of 1.5 gm/kg/day dissolved in water until resolution of fecal impaction or a maximum till 6 days whichever is earlier. Fecal impaction Resolution is defined as passage of clear liquid stool and no palpable abdominal fecolith
  Interventions: Drug: Administration of Polyethylene Glycol (PEG) 3350 + Electrolyte as per treatment allocation to participants
- Polyethylene glycol (PEG) 4000 ARM (Experimental): PEG 4000 will be administered at a dose of 1.5 gm/kg/day dissolved in water until resolution of fecal impaction or a maximum till 6 days whichever is earlier. Fecal impaction Resolution is defined as : Passage of clear liquid stool and no palpable abdominal fecolith
  Interventions: Drug: Administration of Polyethylene Glycol (PEG) 4000 as per treatment allocation to participants

INTERVENTIONS:
Drug: Administration of Polyethylene Glycol (PEG) 4000 as per treatment allocation to participants — As per treatment allocation, PEG 4000 will be administered to participants at a dose of 1.5 gm/kg/day dissolved in water until resolution of fecal impaction or a maximum till 6 days whichever is earlier. Fecal impaction Resolution is defined as : Passage of clear liquid stool and no palpable abdominal fecolith
  Arms: Polyethylene glycol (PEG) 4000 ARM
Drug: Administration of Polyethylene Glycol (PEG) 3350 + Electrolyte as per treatment allocation to participants — As per treatment allocation, PEG 3350 + Electrolytes will be administered to participants at a dose of 1.5 gm/kg/day dissolved in water until resolution of fecal impaction or a maximum till 6 days whichever is earlier. Fecal impaction Resolution is defined as : Passage of clear liquid stool and no palpable abdominal fecolith
  Arms: Polyethylene glycol (PEG) 3350 +Electrolytes ARM

SUMMARY:
Childhood constipation is a common but serious gastrointestinal disorder prevalent worldwide. In 90-95% of children, it is of functional origin. Thirty to seventy-five percent of children with functional constipation also have fecal impaction. The treatment strategy for functional constipation includes fecal disimpaction and maintenance therapy to ensure regular bowel movements.

Polyethylene glycol (PEG) based laxatives have been recommended as the first-line therapeutic agents. The commonly used formulations are PEG 3350 with a molecular weight between 3200- 3700 g/mol and PEG 4000 with molecular weight of 4000 g/mol. Both are shown to be effective in pediatric constipation management in placebo-controlled trials. PEG 3350 + Electrolyte (E) is more widely used than PEG 4000 for the management of constipation. This might be because of the perception that PEG 3350 + E is safer in terms of preventing electrolyte imbalance. However, because of the inclusion of electrolytes, PEG 3350+ E solution taste saltier than PEG 4000. Many patients struggle to tolerate the unpleasant taste resulting in the high incidence of non-compliance. To date, no pediatric trials have compared PEG 4000 versus PEG 3350+E for management of Fecal disimpaction.

Present study has been planned to evaluate the efficacy & tolerability of PEG 4000 versus PEG 3350+ E for fecal disimpaction in pediatric functional constipation. Patients between age 1-16 years having functional constipation (as per ROME IV criteria) with fecal impaction will be included. Subjects will be randomly assigned to either PEG 4000 or PEG 3350+E at a ratio of 1:1. They will be stratified into 3 different age groups: 1-5 years, 6-11 years, and 12-16 years. They will receive either of the PEG solutions (as per allocation) at a dose of 1.5 gm/kg/day for 6 consecutive days or till the resolution of fecal impaction whichever is earlier. The resolution of fecal impaction is defined as the passage of clear liquid stool and the disappearance of palpable abdominal fecolith.

Primary outcome is defined as the proportion of subjects achieving fecal disimpaction in each arm.

Secondary outcomes are defined as follows:

1. Total no of Days required to achieve fecal disimpaction in each arm
2. Cumulative dose of PEG required for fecal disimpaction in each arm
3. Proportion of subjects (> 5 years age) reporting palatability issues in each arm
4. Proportion of subjects discontinuing the treatment due to palatability issues in each arm

DETAILED DESCRIPTION:
Childhood constipation is a common but serious gastrointestinal disorder prevalent worldwide. In approximately 90-95% of children, it is of functional origin i.e., without an identifiable organic pathology. It accounts for 3% of pediatric outpatient visits and 25% of referrals to a pediatric gastroenterologist. Prevalence rates ranging from 0.7% to 29.6% with a median of 8.9% have been described in the older literature, with a higher prevalence in Asian population. However, in a recent study, using the Rome IV criteria, the pooled global prevalence of pediatric functional constipation is found to be 14.4% (95%CI: 11.2-17.6). Severe longstanding constipation is distressing for the entire family and poses a substantial psychological, social, and educational strain on the child's development.

Thirty to seventy-five percent of children with functional constipation also have fecal impaction. It typically begins after several bouts of painful bowel movements, which triggers a vicious cycle of fear-induced stool-withholding behavior leading to more stool retention. Consequently, a significant amount of feces accumulates in the rectum forming a big fecal mass or fecaloma, causing a variety of complaints, including gastrointestinal discomfort, excessive flatulence, nausea or vomiting, poor appetite, mood swings & irritability. European Society for Pediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN) & the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition (NASPGHAN) position paper on pediatric constipation defines fecal impaction as any one of the following: i) palpation of a hard mass in the lower abdomen on physical examination, ii) a dilated rectum filled with a large amount of stool on rectal examination, iii) abdominal radiography showing excessive stool in the distal colon.

The treatment strategy for functional constipation includes fecal disimpaction and maintenance therapy to ensure regular bowel movements. ESPGHAN & NASPGHAN guidelines emphasize that maintenance therapy remains ineffective until disimpaction has been achieved. If initial disimpaction is skipped, oral laxative therapy may paradoxically worsen fecal incontinence/encopresis attributable to overflow diarrhea.

Polyethylene glycol (PEG) based laxatives have been recommended as the first-line therapeutic agents for both disimpaction as well as maintenance therapy in childhood functional constipation. PEG, a biologically inert polymer of the formula H(OCH2CH2)nOH in which n is 68-84. These are non-absorbable polymers, that create an osmotic gradient in the intestinal lumen leading to fluid retention which in turn softens and loosens the stool. Hence, they act as osmotic laxatives. As it does not carry any electrical charge, it does not influence the movement of any other solutes. The commonly used formulations are PEG 3350 with a molecular weight between 3200 and 3700 g/mol and PEG 4000 with an approximate molecular weight of 4000 g/mol. Both are shown to be effective in pediatric constipation management in placebo-controlled trials. However, there is scanty literature available comparing other aspects of various PEG formulations, such as tolerability, palatability, & convenience of administration, which may affect treatment adherence and thus the ultimate treatment outcome. PEG + Electrolyte (E) is more widely used than PEG for the management of constipation. This might be because of the perception that PEG + E is safer in terms of preventing electrolyte imbalance.

However, several head-to-head trials using different PEG formulations in adult constipation patients, showed comparable efficacy and safety. Because of the inclusion of electrolytes, PEG+E tastes saltier than PEG. Many patients struggle to tolerate the unpleasant taste resulting in the high incidence of non-compliance and treatment failure . Two studies from the adult population have demonstrated better acceptance of PEG in comparison to PEG+E . In fact, the latest meta-analysis concluded that the addition of electrolytes to PEG does not provide any clinical benefits over PEG alone.

In a recent double-blind RCT, PEG 4000 is found to be equally efficacious and safe as PEG 3350 + E as a long-term maintenance therapy in children with functional constipation . However, they have not described the tolerability or acceptability data of the cohort. There is only a single pediatric study that showed, PEG 4000 is equally effective and had a higher patient acceptance rate owing to significantly lesser nausea, vomiting episodes, and better palatability compared to PEG 3350. However, both these studies are majorly focused on the comparison between PEG 3350 + E versus PEG 4000 as a long-term maintenance therapy in pediatric functional constipation. There is only a single study that compared PEG 3350 versus PEG 3350 only laxative for fecal disimpaction. Both of them were found to almost equally effective in resolution of fecal impaction, however PEG 3350 + E group had significantly higher side effects as compared to PEG 3350 only laxative.

To date, no pediatric trials have compared PEG versus PEG+E on a head-to-head basis for the treatment of the initial but most important & crucial step of pediatric function constipation management i.e. Fecal disimpaction. Since fecal disimpaction requires administration of a significantly larger volume of PEG administration, palatability becomes a major factor determining the success of disimpaction. On the other hand, there is also of higher possibility of side effects like electrolyte & acid base imbalances because of higher purge rate during disimpaction. Comparison of both these parameters namely tolerability/palatability and safety/side effects profile of PEG versus PEG + E during fecal disimpaction in pediatric population has not been studied previously.

Therefore, the present study has been planned with an aim to evaluate the efficacy & tolerability of PEG 4000 versus PEG 3350+ electrolytes for fecal disimpaction in paediatric functional constipation.

ELIGIBILITY:
Inclusion Criteria:

- 1-16 years age admitted to the inpatient department 2. Having h/o functional constipation as per ROME IV criteria 3)with Fecal impaction defined as A hard mass in the lower abdomen identified on physical examination or Dilated rectum filled with large amount of stool on per rectal Examination or Excessive stool in the colon on abdominal radiography as determined by a radiologist

Exclusion Criteria:

1. Patients with drug-induced constipation
2. Organic constipation ie, I.Neurological disorders eg. Neural tube defects/cerebral/motor neuron diseases/neuro regression syndromes II.Hirschsprung disease, or anal anomalies III.Known metabolic or endocrine disorders
3. Patients with previous gastrointestinal surgery (except appendectomy)
4. Children with suspected gastrointestinal obstruction
5. Patients taking PEG (either at the time of enrolment or within 2 month before enrolment)
6. Patients receiving medication at enrolment or within 1 month before enrolment influencing gastrointestinal motility function (eg, lactulose, loperamide, cisapride)
7. Known history of Allergy to PEG formulations
8. Patients having comorbidity of any other system like CVS/Respiratory/CNS etc
9. Known case of Chronic kidney disease or history of acute kidney injury in past 3 monthes

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving fecal disimpaction in Each Arm | 6 days from allocation of treatment or resolution of fecal impaction whichever is earlier
  The proportion of subjects achieving fecal disimpaction in Each Arm

SECONDARY OUTCOMES:
Total no of Days required to achieve fecal disimpaction in each arm | 6 days from allocation of treatment or resolution of fecal impaction whichever is earlier
  Total no of Days required to achieve fecal disimpaction in each arm
Cumulative PEG dose required for fecal disimpaction in each arm | 6 days from allocation of treatment or resolution of fecal impaction whichever is earlier
  Cumulative PEG dose required for fecal disimpaction in each arm
Proportion of subjects reporting palatability issues in each arm | 6 days from allocation of treatment or resolution of fecal impaction whichever is earlier
  Proportion of subjects reporting palatability issues in each arm
Proportion of subjects discontinuing the treatment due to palatability issues in each arm | 6 days from allocation of treatment or resolution of fecal impaction whichever is earlier
  Proportion of subjects discontinuing the treatment due to palatability issues in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Panda, MD, DM, Principal Investigator — Associate Professor
Locations (1):
- Institute of Medical Sciences (IMS) and SUM Hospital, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benninga MA, Voskuijl WP, Taminiau JA. Childhood constipation: is there new light in the tunnel? J Pediatr Gastroenterol Nutr. 2004 Nov;39(5):448-64. doi: 10.1097/00005176-200411000-00002. No abstract available. PMID 15572881
- [Result] Rubin G, Dale A. Chronic constipation in children. BMJ. 2006 Nov 18;333(7577):1051-5. doi: 10.1136/bmj.39007.760174.47. No abstract available. PMID 17110723
- [Result] van den Berg MM, Benninga MA, Di Lorenzo C. Epidemiology of childhood constipation: a systematic review. Am J Gastroenterol. 2006 Oct;101(10):2401-9. doi: 10.1111/j.1572-0241.2006.00771.x. PMID 17032205
- [Result] Tran DL, Sintusek P. Functional constipation in children: What physicians should know. World J Gastroenterol. 2023 Feb 28;29(8):1261-1288. doi: 10.3748/wjg.v29.i8.1261. PMID 36925458
- [Result] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Result] Shatnawi MS, Alrwalah MM, Ghanma AM, Alqura'an ML, Zreiqat EN, Alzu'bi MM. Lactulose versus polyethylene glycol for disimpaction therapy in constipated children, a randomized controlled study. Sudan J Paediatr. 2019;19(1):31-36. doi: 10.24911/SJP.106-1546805996. PMID 31384086
- [Result] Tabbers MM, DiLorenzo C, Berger MY, Faure C, Langendam MW, Nurko S, Staiano A, Vandenplas Y, Benninga MA; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition; North American Society for Pediatric Gastroenterology. Evaluation and treatment of functional constipation in infants and children: evidence-based recommendations from ESPGHAN and NASPGHAN. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):258-74. doi: 10.1097/MPG.0000000000000266. PMID 24345831
- [Result] Alper A, Pashankar DS. Polyethylene glycol: a game-changer laxative for children. J Pediatr Gastroenterol Nutr. 2013 Aug;57(2):134-40. doi: 10.1097/MPG.0b013e318296404a. PMID 23591910
- [Result] Treepongkaruna S, Simakachorn N, Pienvichit P, Varavithya W, Tongpenyai Y, Garnier P, Mathiex-Fortunet H. A randomised, double-blind study of polyethylene glycol 4000 and lactulose in the treatment of constipation in children. BMC Pediatr. 2014 Jun 19;14:153. doi: 10.1186/1471-2431-14-153. PMID 24943105
- [Result] Candy DC, Edwards D, Geraint M. Treatment of faecal impaction with polyethelene glycol plus electrolytes (PGE + E) followed by a double-blind comparison of PEG + E versus lactulose as maintenance therapy. J Pediatr Gastroenterol Nutr. 2006 Jul;43(1):65-70. doi: 10.1097/01.mpg.0000228097.58960.e6. PMID 16819379
- [Result] Youssef NN, Peters JM, Henderson W, Shultz-Peters S, Lockhart DK, Di Lorenzo C. Dose response of PEG 3350 for the treatment of childhood fecal impaction. J Pediatr. 2002 Sep;141(3):410-4. doi: 10.1067/mpd.2002.126603. PMID 12219064
- [Result] Bekkali NL, van den Berg MM, Dijkgraaf MG, van Wijk MP, Bongers ME, Liem O, Benninga MA. Rectal fecal impaction treatment in childhood constipation: enemas versus high doses oral PEG. Pediatrics. 2009 Dec;124(6):e1108-15. doi: 10.1542/peds.2009-0022. PMID 19948614
- [Result] Miller MK, Dowd MD, Friesen CA, Walsh-Kelly CM. A randomized trial of enema versus polyethylene glycol 3350 for fecal disimpaction in children presenting to an emergency department. Pediatr Emerg Care. 2012 Feb;28(2):115-9. doi: 10.1097/PEC.0b013e3182442c0a. PMID 22270500
- [Result] Seinela L, Sairanen U, Laine T, Kurl S, Pettersson T, Happonen P. Comparison of polyethylene glycol with and without electrolytes in the treatment of constipation in elderly institutionalized patients: a randomized, double-blind, parallel-group study. Drugs Aging. 2009;26(8):703-13. doi: 10.2165/11316470-000000000-00000. PMID 19685935
- [Result] Chaussade S, Minic M. Comparison of efficacy and safety of two doses of two different polyethylene glycol-based laxatives in the treatment of constipation. Aliment Pharmacol Ther. 2003 Jan;17(1):165-72. doi: 10.1046/j.1365-2036.2003.01390.x. PMID 12492746
- [Result] Szojda MM, Mulder CJ, Felt-Bersma RJ. Differences in taste between two polyethylene glycol preparations. J Gastrointestin Liver Dis. 2007 Dec;16(4):379-81. PMID 18193118
- [Result] Katelaris P, Naganathan V, Liu K, Krassas G, Gullotta J. Comparison of the effectiveness of polyethylene glycol with and without electrolytes in constipation: a systematic review and network meta-analysis. BMC Gastroenterol. 2016 Mar 31;16:42. doi: 10.1186/s12876-016-0457-9. PMID 27029340
- [Result] Bekkali NLH, Hoekman DR, Liem O, Bongers MEJ, van Wijk MP, Zegers B, Pelleboer RA, Verwijs W, Koot BGP, Voropaiev M, Benninga MA. Polyethylene Glycol 3350 With Electrolytes Versus Polyethylene Glycol 4000 for Constipation: A Randomized, Controlled Trial. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):10-15. doi: 10.1097/MPG.0000000000001726. PMID 28906317
- [Result] Savino F, Viola S, Erasmo M, Di Nardo G, Oliva S, Cucchiara S. Efficacy and tolerability of peg-only laxative on faecal impaction and chronic constipation in children. A controlled double blind randomized study vs a standard peg-electrolyte laxative. BMC Pediatr. 2012 Nov 15;12:178. doi: 10.1186/1471-2431-12-178. PMID 23152962
- [Result] Boles EE, Gaines CL, Tillman EM. Comparison of Polyethylene Glycol-Electrolyte Solution vs Polyethylene Glycol-3350 for the Treatment of Fecal Impaction in Pediatric Patients. J Pediatr Pharmacol Ther. 2015 May-Jun;20(3):210-6. doi: 10.5863/1551-6776-20.3.210. PMID 26170773